CLINICAL TRIAL: NCT00628381
Title: Arginine and Nitric Oxide (NO) Metabolism in Sepsis; L-citrulline Enteral Supplementation for the Normalisation of the Arginine-NO Metabolism
Brief Title: L-citrulline Supplementation During Sepsis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: M.Poeze, MD, PhD,, Department of surgery, University hospital Maastricht
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEC-08; ZON/NW 40-00806-98-114
Record Dates: First submitted 2008-02-26; First posted 2008-03-05 (Estimated); Last update posted 2010-09-03 (Estimated); Status verified 2010-09

CONDITIONS: Sepsis; Multiple Organ Failure
Keywords: sepsis; microcirculation; nitric oxide; citrulline
MeSH Terms: conditions — Sepsis; Multiple Organ Failure | interventions — Alanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AA (Experimental): 24 ICU patients with severe sepsis will get a L-citrulline 8 h enteral supplementation.
  Interventions: Dietary Supplement: L-citrulline supplementation
- AB (Active Comparator): 24 ICU patients with severe sepsis will get an alternative isocaloric amino acid supplementation (L-alanine) during 8 hours
  Interventions: Dietary Supplement: L-alanine

INTERVENTIONS:
Dietary Supplement: L-citrulline supplementation — L-citrulline, 1.8micromol/kg/min, during 8 hours continuously supplemented
  Arms: AA
Dietary Supplement: L-alanine — L-alanine enteral infusion, isocaloric dosage (3.6 micromol/kg/min), during 8 hours, continuously supplemented
  Arms: AB

SUMMARY:
The purpose of this study is to study the stimulating effects of prolonged (8h) enteral L-citrulline supplementation on the normalisation of the plasma citrulline concentrations and the Arginine-NO metabolism, the microcirculation, the systemic hemodynamics, vascular permeability, and organ function and disease severity scores.

DETAILED DESCRIPTION:
NO synthesis is compromised during sepsis through lack of arginine de novo synthesis and may thereby contribute to impaired microcirculation and organ dysfunction. Supplementation of L-citrulline in septic patients will increase NO production without increased arginase activity and these effects will be studied on arginine-NO metabolism,improved organ function, vascular permeability and microcirculation.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from close relative
* Age > 18 years
* Patient meets the general criteria for severe sepsis or septic shock, diagnosed less than 48 h prior to study inclusion.
* Patient must be relatively hemodynamically stable, defined as stable blood pressure (variation in mean arterial pressure <15 mm Hg) during 2h without necessity of increasing the vasopressor dose, inotropic support or rate of fluid administration.
* Systemic arterial catheter in place with continuous pressure monitoring.
* Patients in whom the clinician is prepared to provide full life support during the duration of the study

Exclusion Criteria:

* Shock due to any cause other than sepsis (e.g. drug reaction or drug overdose, pulmonary embolus, burn injury etc.)
* Prolonged or high dose corticosteroid use
* Liver cirrhosis
* Chronic pancreatitis
* Insulin-dependent diabetes mellitus
* Metastases, haematological malignancies or chemotherapy
* Patients on dialysis (CVVH or other)
* Pre-existent renal failure (on dialysis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
To study stimulating effects of prolonged (8h) enteral L-citrulline supplementation on the normalisation of the arginine-NO metabolism | 8 hours

SECONDARY OUTCOMES:
Secondary study endpoints are the microcirculation, the vascular permeability and organ function scores. | within 8 hours

CONTACTS AND LOCATIONS:
Overall Officials: Martijn Poeze, MD, PhD, Principal Investigator — Department of Surgery
Locations (1):
- University Hospital Maastricht, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Rouge C, Des Robert C, Robins A, Le Bacquer O, Volteau C, De La Cochetiere MF, Darmaun D. Manipulation of citrulline availability in humans. Am J Physiol Gastrointest Liver Physiol. 2007 Nov;293(5):G1061-7. doi: 10.1152/ajpgi.00289.2007. Epub 2007 Sep 27. PMID 17901164
- [Background] Barr FE, Tirona RG, Taylor MB, Rice G, Arnold J, Cunningham G, Smith HA, Campbell A, Canter JA, Christian KG, Drinkwater DC, Scholl F, Kavanaugh-McHugh A, Summar ML. Pharmacokinetics and safety of intravenously administered citrulline in children undergoing congenital heart surgery: potential therapy for postoperative pulmonary hypertension. J Thorac Cardiovasc Surg. 2007 Aug;134(2):319-26. doi: 10.1016/j.jtcvs.2007.02.043. PMID 17662768
- [Background] Lehr HA, Bittinger F, Kirkpatrick CJ. Microcirculatory dysfunction in sepsis: a pathogenetic basis for therapy? J Pathol. 2000 Feb;190(3):373-86. doi: 10.1002/(SICI)1096-9896(200002)190:33.0.CO;2-3. PMID 10685071
- [Background] Wu G, Morris SM Jr. Arginine metabolism: nitric oxide and beyond. Biochem J. 1998 Nov 15;336 ( Pt 1)(Pt 1):1-17. doi: 10.1042/bj3360001. PMID 9806879
- [Background] Hallemeesch MM, Lamers WH, Deutz NE. Reduced arginine availability and nitric oxide production. Clin Nutr. 2002 Aug;21(4):273-9. doi: 10.1054/clnu.2002.0571. PMID 12135586